CLINICAL TRIAL: NCT03321344
Title: Safety and Initial Feasibility of Using the Neurolyser XR Device for the Treatment of Facet Related Low Back Pain
Brief Title: Safety and Initial Feasibility of Using the Neurolyser for Facet Related Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FUSMobile Inc. (Industry)
Collaborators: Focused Ultrasound Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LBP-001
Record Dates: First submitted 2017-10-18; First posted 2017-10-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2020-07

CONDITIONS: Facet Related Low Back Pain

STUDY DESIGN:
Intervention Model Description: Single arm, non-randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test Arm (Experimental): Focused Ultrasound Thermal ablation of the Medial Nerve Branch
  Interventions: Device: Focused Ultrasound Thermal ablation

INTERVENTIONS:
Device: Focused Ultrasound Thermal ablation — Focused Ultrasound Thermal ablation of the Medial Nerve Branch

SUMMARY:
Single arm pilot study to evaluate the safety and initial feasibility of the Neurolyser XR, a new portable high intensity focused ultrasound device, for noninvasive thermal ablation of medial nerve branches of painful lumbar facet joint/s

DETAILED DESCRIPTION:
Study design: Prospective, single arm

Timeline: six month enrollment period and 12 months follow-up period.

Sites: The study will be conducted at McGill University.

Study population: Ten adult patients diagnosed with facet related low back pain.

Primary study objective: Safety and efficacy of the Neurolyser XR for the treatment of facet related low back pain.

Safety would be evaluated by the incidence and severity of treatment related adverse events Efficacy would be evaluated by the changes in average pain score and Rolland Morris Disability Questionnaire between baseline and 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and females, legally able and willing to participate in the study and come for follow-up visits
2. Able and willing to fill the study forms and to communicate with investigator
3. Patient with uni or bilateral lumbar facetogenic pain of > 6 months duration
4. Patients presenting with a) a positive (>70% pain relief) to a previous L1 to L5 lumbar medial branch block and / or b) with a positive (>70% pain relief) to a previous lumbar facet thermal RF denervation within the last 6 months)
5. Average pain score of 4 or higher in the last month, (on a scale of 0 to 10)

Exclusion Criteria:

1. Pregnant or breastfeeding patient
2. Patients younger than 18 or older than 80 years
3. Patients presenting with neurological deficits (including lumbosacral radiculopathy but not radicular pain).
4. History of spine surgery
5. Presence of metal hardware at the lumbosacral spine
6. Lumbar spine pathology that may increase procedural risk and / or influence symptoms and / or generate unrelated adverse event, (per the discretion of the study PI)
7. Patients unable to understand and complete the research questionnaires in English or French
8. Any severe medical condition preventing the patient from safely and effectively being treated in the study or reporting study outcome.
9. Patient with extensive scarring in the skin and tissue overlying the treatment area.
10. Patients enrolled in or planned to be enrolled in another clinical trial during the duration of this research project

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
NRS | Base line, 2 days 1, 2 & 4 weeks, 3, 6 & 12 months after procedure
  Reduction in average pain score as measured by a numeric rating scale from 0 (no pain) to 10, worst possible pain
RMD | Base line, 1 & 4 weeks, 3, 6 & 12 months after procedure
  Reduction in Rolland Morris Disability Questionnaire score
Saftey | Base line, Procedure day, 2 days 1, 2 & 4 weeks, 3, 6 & 12 months after procedure
  Safety will be measured by the incidence and severity of treatment related adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Alan Edwards Pain Management Unit - Montreal General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perez J, Gofeld M, Leblang S, Hananel A, Aginsky R, Chen J, Aubry JF, Shir Y. Fluoroscopy-Guided High-Intensity Focused Ultrasound Neurotomy of the Lumbar Zygapophyseal Joints: A Clinical Pilot Study. Pain Med. 2022 Jan 3;23(1):67-75. doi: 10.1093/pm/pnab275. PMID 34534337